CLINICAL TRIAL: NCT05014867
Title: A Prospective, Four Arms, Open Label, Comparative Study to Assess the Ongoing Pregnancy Rate for Poor Responders Women Undergoing Different Embryo Transfer Protocols
Brief Title: Comparative Study to Assess the Ongoing Pregnancy Rate for Poor Responders Women Undergoing Different Embryo Transfer Protocols
Status: Completed | Type: Observational
Sponsor: Wael Elbanna Clinic (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Wael Elbanna, Managing director for Wael Elbanna Clinic, Wael Elbanna Clinic
Other Study IDs: Elbanna_003
Record Dates: First submitted 2021-08-14; First posted 2021-08-20 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Embryo Transfer in Poor Responders
Keywords: Poor responders; PGS; Sequential; Embryo transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Arm 1: Poor responders women undergoing frozen sequential embryo transfer on Day 3 and Day 5
  Interventions: Procedure: Embryo transfer method
- Arm 2: Poor responders women undergoing sequential fresh embryo transfer on Day 3 and Day 5
  Interventions: Procedure: Embryo transfer method
- Arm 3: Poor responders women undergoing sequential embryo transfer on Day 3 and Day 5 after performing PGS
  Interventions: Procedure: Embryo transfer method
- Arm 4: Poor responders women undergoing conventional frozen embryo transfer on Day 5
  Interventions: Procedure: Embryo transfer method

INTERVENTIONS:
Procedure: Embryo transfer method — 1. Sequential embryo transfer on day 3 and day 5 in a frozen cycle
  2. Sequential embryo transfer on day 3 and day 5 in a fresh cycle
  3. Sequential embryo transfer on day 3 and day 5 after performing PGS
  4. Conventional Day 5 frozen embryo transfer

SUMMARY:
Published data on sequential transfer are limited and are not consistent. Also, further research into methods of risk combination and assessment, would allow us to help our patients make better-informed decisions about whether or not to proceed with invasive diagnostic tests as the PGS. So our study aims to describe the ongoing pregnancy rate for poor responders women undergoing four different embryo transfer protocols among four arms within the study. Moreover, to describe the miscarriage rate, and the baseline characteristics for the same population. This clinical study will be conducted in compliance with the clinical study protocol and applicable regulatory requirements.

DETAILED DESCRIPTION:
The study aims to describe the ongoing pregnancy rate for poor responders women undergoing four different embryo transfer protocols among four arms within the study. Moreover, to describe the miscarriage rate, and the baseline characteristics for the same population. This clinical study will be conducted in compliance with the clinical study protocol and applicable regulatory requirements.

This study is prospective, comparative, open label and multi-center study. The study participants' relevant medical records will be collected and reviewed after obtaining informed consent for the participants.

The study materials that will be used will include blood tests, and ultrasound. The study will involve four study arms:

Arm 1: Poor responders women undergoing frozen sequential embryo transfer on Day 3 and Day 5 Arm 2: Poor responders women undergoing sequential fresh embryo transfer on Day 3 and Day 5 Arm 3: Poor responders women undergoing sequential embryo transfer on Day 3 and Day 5 after performing PGS Arm 4: Poor responders women undergoing conventional frozen embryo transfer on Day 5

Primary and secondary key measurements will be used in the study.

The primary measures will include:

* Presence of intrauterine gestational sac at 12 weeks beyond embryo transfer
* Presence of fetal heart pulsation at 12 weeks beyond embryo transfer

The secondary key measures will include:

* Occurance of abortion between week 7 and week 20 of gestation
* Recording the the baseline characteristics of the study participants

ELIGIBILITY:
Inclusion Criteria:

1. The age group of these women is 25-45 years
2. Normal endometrial cavity confirmed by hysteroscopy
3. Poor responders with AMH <1
4. Patients with at least grade 1 days 3 embryo and grade 1 day 5 frozen embryos

Exclusion Criteria:

1. Patients with any immunological disorders
2. Patients with uncontrolled systemic diseases
3. Patients with previous uterine surgeries except for Cesarean section

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Poor responders women undergoing one of the following:
  1. Sequential embryo transfer on day 3 and day 5 in a frozen cycle
  2. Sequential embryo transfer on day 3 and day 5 in a fresh cycle
  3. Sequential embryo transfer on day 3 and day 5 after performing PGS
  4. Conventional Day 5 frozen embryo transfer
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy rate for poor responders women in the four arms | Till the end of 12 weeks of gestation
  Recording the following for the four arms of the study:
  * Presence of intrauterine gestational sac at 12 weeks beyond embryo transfer
  * Presence of fetal heart pulsation at 12 weeks beyond embryo transfer

SECONDARY OUTCOMES:
miscarriage rate for poor responders women in the four arms | Till the end of 20 weeks of gestation
  Recording the following for the four arms of the study:
  - Occurance of abortion between week 7 and week 20 of gestation
The baseline characteristics of the study participants | Before study intervention of the four arms (at day 2 in the ovulation induction cycle)
  Recording the following for the four arms of the study:
  -age , body mass index in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Wael Elbanna Clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided